CLINICAL TRIAL: NCT02615405
Title: Phospholipid Hypothesis of Depression: From Molecular Biology, Neuroimaging to Behaviour
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, Kuan-Pin, China Medical University Hospital, National Science and Technology Council, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NSC101-2628-B-039-001-MY3
Record Dates: First submitted 2015-11-24; First posted 2015-11-26 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-11

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- EPA (Experimental): 3.5 g/day in Studies 1 & 2
  Interventions: Dietary Supplement: EPA
- DHA (Active Comparator): 1.75 g/day in Studies 1 & 2
  Interventions: Dietary Supplement: DHA
- Placebo capsules (Placebo Comparator): oleic oil in Study 1
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: EPA — A daily treatment of 5 identical capsules of EPA (3.5 g/d) for Studies 1 & 2.
  Other Names: Fish oil EPA
  Arms: EPA
Dietary Supplement: DHA — A daily treatment of 5 identical capsules of DHA (1.75 g/d) for Studies 1 & 2.
  Other Names: Fish oil DHA
  Arms: DHA
Dietary Supplement: Placebo — A daily treatment of 5 identical capsules of placebo (high oleic oil) in single or divided administration for Study 1.
  Other Names: oleic oil
  Arms: Placebo capsules

SUMMARY:
With the dissatisfaction of monoamine-based pharmacotherapy and the high comorbidity of physical illness in depression, the serotonin hypothesis seems to fail in approaching the etiology of depression. Based upon the evidence from epidemiological data, case-control studies of PUFAs compositions, and antidepressant effects in clinical trials, phospholipid polyunsaturated fatty acids (PUFAs) is enlightening a promising path to discover the unsolved of depression.

DETAILED DESCRIPTION:
There are several important questions to answer regarding phospholipid polyunsaturated fatty acids (PUFAs) hypothesis of depression. Firstly, although case-control studies revealed that depressive patients had lower levels of omega-3 PUFAs, the abnormal findings in individual PUFA of docosahexaenoic acid (DHA), eicosapentaenoic acid (EPA) or arachidonic acid (AA) are not consistent. Secondly, the deficits in n-3 PUFAs are related to their metabolic enzymes. However, the association study of polymorphisms of PUFA-metabolism related genes in depression is limited. Thirdly, the active component of antidepressant effect in n-3 PUFAs is still in debate. Fourthly, the molecular mechanisms of n-3 PUFAs' antidepressant effects have yet to be elucidated in human brain functional neuroimaging or in cellular models.

This 3-year proposal is divided into 2 clinical studies. In study 1, the investigators aim to test the clinical and biological effects of n-3 PUFAs (EPA: 3.5 g/d and DHA: 1.75 g/d versus placebo: high oleic oil) for depressive symptoms in a 12-week, double-blind, placebo-controlled trial of patients with drug-free MDD. In study 2, the investigators will measure the biological and neuroimaging markers to investigate the biological mechanisms of EPA (3.5 g/d) versus DHA (1.75 g/d) in 12-week, double-blind, randomized-controlled trial with patients with drug-free major depression disorder (MDD).

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic and Statistical Manual (DSM)-IV criteria for major depressive disorder
* Age being age 18-65.
* Capacity and willingness to give written informed consent.
* Free from antidepressants, mood stabilizers, and antipsychotics for more than 4 weeks.

Exclusion Criteria:

* Any major medical illnesses.
* A recent or past history of any Axis-I diagnoses besides major depressive disorder, including psychotic disorders; cognitively impaired mental disorders; impulse control disorders; substance use disorder or substance abuse (last 6 months prior to the studies); primary anxiety disorders, including post-traumatic stress disorder and panic disorder; and bipolar disorders; or Axis-II diagnoses, i.e. borderline and antisocial personality disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2012-08; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Changes from Baseline Hamilton Depression Rating Scale (HDRS) at 12 weeks | Week 12
Remission rate | Week 12
Response rate | Week 12

SECONDARY OUTCOMES:
Changes in Beck Depression Inventory (BDI) | Week 12
Changes in Neurotoxicity Rating Scale (NRS) | Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Kuan-Pin Su, MD PhD, Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan, Taiwan

REFERENCES:
- [Derived] Su KP, Yang HT, Chang JP, Shih YH, Guu TW, Kumaran SS, Galecki P, Walczewska A, Pariante CM. Eicosapentaenoic and docosahexaenoic acids have different effects on peripheral phospholipase A2 gene expressions in acute depressed patients. Prog Neuropsychopharmacol Biol Psychiatry. 2018 Jan 3;80(Pt C):227-233. doi: 10.1016/j.pnpbp.2017.06.020. Epub 2017 Jun 23. PMID 28648567